CLINICAL TRIAL: NCT06045793
Title: A Single-Blind, Randomized Study Comparing The Efficacy And Safety Of A Single Dose Of TNX-1300 To Placebo With Usual Care For The Treatment Of Signs And Symptoms Of Acute Cocaine Intoxication In Emergency Department Subjects (CATALYST Study)
Brief Title: Comparing Efficacy & Safety Of TNX-1300 To Placebo With UC For Treatment Of Acute Cocaine Intoxication In ED Subjects (CATALYST)
Acronym: CATALYST
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Tonix has discontinued enrollment and terminated the Phase 2 CATALYST study (TNX-CE-CI202) because enrollment in this emergency department-based study was slower than projected. The study was not discontinued for safety or efficacy reasons.
Sponsor: Tonix Pharmaceuticals, Inc. (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Premier (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TNX-CE-CI202; 5U01DA056245 (NIH)
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Cocaine Use; Cocaine Intoxication; Cocaine Toxicity; Cocaine Abuse; Cocaine Adverse Reaction
Keywords: Emergency Department; Cocaine; Cocaine Intoxication; Cocaine Esterase
MeSH Terms: conditions — Cocaine-Related Disorders; Emergencies | interventions — Injections; cocaine esterase

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients will be blinded to which treatment arm they are assigned to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- TNX-1300 (Experimental): A single IV 200 mg injection of TNX-1300
  Interventions: Drug: TNX-1300 (Injection)
- Placebo (Placebo Comparator): A single IV injection of placebo with UC
  Interventions: Drug: Placebo (Injection)

INTERVENTIONS:
Drug: TNX-1300 (Injection) — Patients will receive a single IV injection of TNX-1300.
  Other Names: Cocaine esterase
  Arms: TNX-1300
Drug: Placebo (Injection) — Patients will receive a single IV injection of placebo with usual care (UC).
  Arms: Placebo

SUMMARY:
This is a Phase 2 single-blind, randomized, multicenter study to compare the efficacy and safety of a single dose of TNX-1300 to placebo with usual care in patients with acute cocaine intoxication within the emergency department setting.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female and is 18-64 years of age.
* Subject has the capacity to provide voluntary written informed consent. In cases in which the investigator is unclear if the subject has the capacity to consent, a determination regarding capacity must be made by a psychiatrist trained in assessment of capacity to consent to research in order for the subject to be eligible.
* At Screening, subject presents with cardiac symptoms while intoxicated with cocaine, inclusive of elevated systolic or diastolic BP, as defined below, with or without behavioral symptoms:

  * Systolic BP >140 mmHg, or
  * Diastolic BP >90 mmHg Note: subjects with a QT interval corrected for heart rate (QTc) >500 msec may be eligible for study participation, based on investigator judgment.
* At Screening and Baseline assessments, subject must have a SIS total score of ≥4
* At Baseline, subject has a CGI-S score ≥3.
* Subject has a positive urine drug screen test at Pre-screening to confirm cocaine use and detect polysubstance abuse (subject may test positive for cannabinoids and/or opioids and remain eligible; subject may test positive for alcohol by breathalyzer and remain eligible).
* Subject must be willing to practice the following:

  * If female, practice one of the following methods of birth control throughout the study and for 28 days after study drug administration:
  * Hormonal methods such as oral, implantable, injectable, or transdermal contraceptives for a minimum of one full cycle (based on the patient's usual menstrual cycle period) before study drug administration;
  * Intrauterine device;
  * Bilateral tubal ligation
  * Double-barrier method (condoms, sponge, diaphragm, or vaginal ring with spermicidal jelly or cream);
  * If male, practice double-barrier method throughout the study and for 28 days after study drug administration, if female partner is not following birth control methods a-c mentioned above
* Subject is a suitable candidate for investigational treatment based on the opinion of the investigator.

Exclusion Criteria:

* Subject who has been admitted to the ED involuntarily.
* Subject who participated in this clinical study previously.
* Subject has a score of 3 on the systolic and/or diastolic BP SIS components, a "mental state" or "orientation" SIS component score of ≥2, or an "orientation" SIS component score of ≥1 and the subject is not oriented to either person or place (i.e., only disorientation to time is allowed).
* Subject who, at Screening, expresses C-SSRS suicidal ideation of Type 4 or 5 in the prior week or any C-SSRS suicidal behavior in the prior week.
* Subject tests positive for stimulant drugs of abuse other than cocaine, including methylphenidate, 3,4-methylenedioxymethamphetamine, methamphetamine, or other amphetamines at Screening.
* Subject has a clinically significant untreated cardiac condition, such as prior myocardial infarction, current ischemia assessed by ECG-based criteria, aortic dissection, ventricular fibrillation, Torsade de pointes, ventricular tachycardia, cardiomyopathy, pulmonary edema, cardiac arrest, significant conduction disturbance (e.g., greater than first degree heart block), QRS interval >120 msec, or severe or life-threatening hypertension. Untreated hypertension may be allowed if not considered severe or life-threatening. Note: hypertension will be considered severe or life-threatening if systolic BP is >200 mmHg and/or diastolic BP is >130 mmHg.
* Subject incurred or is likely to incur a myocardial infarction or other life-threatening severe event or has acute ECG changes indicative of acute coronary syndrome according to investigator judgment. Such changes may include new, transient, or dynamic ST-segment elevation, ST-depression, or significant Q waves. Based on investigator judgement, T-wave inversion and T-wave flattening may also be considered in the risk assessment for acute coronary syndrome.
* Subject has a heart rate ≥180 bpm, atrial fibrillation, greater than first degree heart block, or chest pain with ECG-based evidence of ischemia.
* Subject has a clinically significant or unstable medical illness, condition, or disorder that can compromise subject safety or adversely affect the evaluation of clinical outcome parameters.
* Subject has a clinical history of anaphylaxis, severe asthma, hypersensitivity, or angioedema.
* Subject requires physical restraints due to physiological and/or behavioral symptoms.
* Subject receives anti-hypertensive medication(s) in the ED prior to study enrollment.
* Subject is pregnant or breastfeeding.
* Participation in another investigational drug study (current or within 30 days of Screening) or previous participation in a study of TNX-1300.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2024-08-16 (Actual); Primary Completion 2025-04-21 (Actual); Study Completion 2025-04-21 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Systolic BP at 60 minutes after dosing, comparing TNX-1300 to placebo with UC | 60 minutes after IV administration
  Patients will undergo a Systolic BP assessment at Baseline and at 60 minutes after dosing.

SECONDARY OUTCOMES:
Change from Baseline in QT interval corrected for heart rate (QTc) at 15 minutes after dosing, comparing TNX-1300 to placebo with UC | 15 minutes after IV administration
  Patients will undergo a 12-lead ECG at Baseline and at 15 minutes after dosing.
Change from Baseline in diastolic BP at 60 minutes after dosing, comparing TNX-1300 to placebo with UC | 60 minutes after IV administration
  Patients will undergo a Diastolic BP assessment at Baseline and at 60 minutes after dosing
Change from Baseline in Stimulant Intoxication Scale (SIS) total score at 60 minutes after dosing, comparing TNX-1300 to placebo with UC | 60 minutes after IV administration
  Patients will be assessed with the SIS for characterizing severity of cocaine intoxication at Baseline and at 60 minutes after dosing. The SIS has 6 items, each of which is scored on a range of 0-3 (4 items) or 0-4 (2 items). The SIS has a total score range of 0 to 20, with 0 being the lowest severity and 20 being the highest severity.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Sullivan, MD, Study Director — Tonix Pharmaceuticals
Locations (6):
- United States (6):
  - University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - University Of Maryland Medical Center, Baltimore, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Wayne State University, Detroit, Michigan
  - Washington University, St Louis, Missouri
  - Baylor College of Medicine, Ben Taub Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No